CLINICAL TRIAL: NCT02104960
Title: Study of Skin Parameters in the PROOF Cohort
Acronym: PEAU PROOF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1308003; 2013-A00094-41 (Other: ANSM)
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Skin Aging
Keywords: Skin Surface Microscopy; Skin Aging; PROOF
MeSH Terms: interventions — Biopsy; Microscopy, Confocal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROOF: Healthy inhabitants of the city of Saint-Etienne, France, and aged 65 years at the inclusion date. (NCT00759304)
  Interventions: Other: Dermatological clinical examination; Other: Biopsy; Other: Confocal microscopy in vivo

INTERVENTIONS:
Other: Dermatological clinical examination — Clinical pictures, Dermatoscopy, Elastography, Sebumetry
Other: Biopsy — Skin biopsy for examinations by confocal microscopy ex vivo and histopathology
Other: Confocal microscopy in vivo — Examination by confocal microscopy in vivo

SUMMARY:
This study aims to evaluate skin aging of an homogeneous population of 77 years old patient selected among the PROOF cohort who has been continuously investigated by cardiological examination.

Skin aging will be explored by macroscopic and microscopic evaluation. In particular, skin aging will be measured by an index of clinical aging (SCINEXA) and other complementary measures such as facial photos, standard and High Definition dermoscopy, elastography, sebumetry, in vivo and ex vivo confocal microscopy, and classical histological examinations.

ELIGIBILITY:
Inclusion Criteria:

* included in the PROOF cohort
* Form consent signed

Exclusion Criteria:

* Past history of surgery and / or treatment of aesthetic medicine
* neurological disorders
* insulin-dependent diabetes,
* corticosteroids or retinoids (isotretinoin, ...) > 1 year

Ages: 75 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: PROOF cohort (NCT00759304)
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
SCINEXA score | Day 1
  The aging of the skin is evaluated by a semi-quantitative composite of 19 clinical variables : the score SCINEXA

SECONDARY OUTCOMES:
in vivo confocal microscopy | Day 1
  Skin aging evaluated by in vivo confocal microscopy
ex vivo confocal microscopy | Day 1
  Skin aging evaluated by ex vivo confocal microscopy ( thickness of the epidermis with and without the stratum corneum, dermis thickness , number of sweat glands per unit volume).
histology | Day 1
  Skin aging evaluated by conventional histology (thickness of the epidermis and dermis, presence and degree of elastosis , flattening of the dermo- epidermal junction)
RAMAN | Day 1
  The composition of subcutaneous fat measured by ex vivo RAMAN spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Elisa CINOTTI, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France